CLINICAL TRIAL: NCT06082245
Title: Comparison Perioperative Analgesia Efficacy Between Thoracolumbar Interfascial Plane Block and Erector Spinae Plane Block for Patients With Lumbar Spine Fusion Surgery: A Randomized Controlled Study
Brief Title: TLIP Block and ESP Block For Perioperative Analgesia In Patients With Lumbar Spine Fusion Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanoi Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HMU10.2023
Record Dates: First submitted 2023-09-26; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-09

CONDITIONS: Analgesia; Spine Fusion
Keywords: perioperation; Thoracolumbar interfasial plane; erector spine plane; ultrasound-guided analgesia; patient-controlled analgesia
MeSH Terms: conditions — Agnosia | interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: TLIP block group, ESP block group and control group
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TLIP Group (Active Comparator): Patients were anesthetized before surgery using TLIP lumbar block (L3) under ultrasound with 20ml of ropivacaine 0.25% anesthetic on each side. After that, the patient was given general anesthesia for surgery
  Interventions: Procedure: TLIP Block For Perioperative Analgesia In Patients With Lumbar Spine Fusion Surgery
- ESP Group (Active Comparator): Patients were anesthetized before surgery with lumbar (L3) ESP block method under ultrasound with 20ml of Ropivacaine 0.25% anesthetic on each side. After that, the patient was given general anesthesia for surgery.
  Interventions: Procedure: ESP Block For Perioperative Analgesia In Patients With Lumbar Spine Fusion Surgery
- Control Group (Experimental): Patients received general anesthesia, then the incision was anesthetized with 15ml of 1% lidocaine mixed with 1/200,000 adrenaline on each side before surgery
  Interventions: Procedure: Lidocaine injection

INTERVENTIONS:
Procedure: TLIP Block For Perioperative Analgesia In Patients With Lumbar Spine Fusion Surgery — * Patients were placed in a prone position;
  * ultrasound-guided TLIP block: (1) The transducer was positioned in a transverse midline position at the level of the L3 vertebra. After the identification of the spinous process and interspinous muscles. (2) The probe was moved laterally to identify the multifidus (MF) and longissimus (LG) muscles. (3) the TLIP block was performed under real-time ultrasound guidance using an insulated 100-mm 22G echogenic needle which was inserted in-plane lateral to the medial direction. (4) After negative aspiration, 20-mL 0.25% ropivacaine was injected in each side bilaterally in the interface between the MF and LG muscles.
  * patients received general anesthesia
  Arms: TLIP Group
Procedure: ESP Block For Perioperative Analgesia In Patients With Lumbar Spine Fusion Surgery — * Patients were placed in a prone position;
  * ultrasound-guided ESP block: (1) The 12th rib was identified in the parasagittal plane, and with probe shifted caudad and medial, the L3 transverse process (TP) was identified. (2) Insulated 100-mm 22G echogenic needle was inserted from cranial to caudal direction. (3) The needle tip was identified between the L2 and L3, and 20 mL of 0.25% ropivacaine was injected in each side bilaterally in ESP.
  * patients received general anesthesia
  Arms: ESP Group
Procedure: Lidocaine injection — * patients received general anesthesia
  * the expected incision was anesthetized with 15ml of 1% lidocaine mixed with 1/200,000 adrenaline on each side before surgery.
  Arms: Control Group

SUMMARY:
Background: Pain relief for lumbar spine surgery is being updated to help improve the quality of post-operative recovery, especially ultrasound-guided pain relief anesthesia methods, including two anesthesia methods. Thoracolumbar interfascial plane block (TLIP block) and erector spinae plane block (ESP block) are increasingly commonly applied. Objective: compare the pain relief effectiveness of TLIP block with ESP block for lumbar spine surgery.

Methods: Randomized prospective intervention study conducted at Hanoi Medical University Hospital from October 2021 to October 2022 including 100 lumbar spine surgery patients randomly divided into three groups: group control, TLIP group and ESP group. Outcomes regarding perioperative pain score (ANIm, VAS), the effectiveness of 2 ultrasound-guided methods, the complications and the side effects were recorded.

DETAILED DESCRIPTION:
* All research patients were divided into 3 groups by random drawing: control group, TLIP group and ESP group.
* TLIP group: patients were anesthetized before surgery using TLIP lumbar block (L3) under ultrasound with 20ml of ropivacaine 0.25% anesthetic on each side. After that, the patient was given endotracheal anesthesia for surgery.
* ESP group: patients were anesthetized before surgery with lumbar (L3) ESP block method under ultrasound with 20ml of Ropivacaine 0.25% anesthetic on each side. After that, the patient was given endotracheal anesthesia for surgery.
* Control group: patients received regular endotracheal anesthesia, then the incision was anesthetized with 15ml of 1% lidocaine mixed with 1/200,000 adrenaline on each side before surgery.
* Anesthesia and monitoring process: all patients in all 3 groups were anesthetized using general anesthesia:

  * Install monitoring to monitor pulse parameters, blood pressure, SpO2, EtCO2.
  * Install an Analgesia Nociception Index (ANI) meter and monitor the ANI index continuously during surgery. Monitor ANI monitor V2 during surgery, maintain ANIm within the range of 50-70.
  * Induction of anesthesia: fentanyl 2mcg/kg slow intravenous injection, wait 3 minutes then inject propofol 2-3mg/kg, rocuronium 0.6mg/kg (when eyelid reflex is lost). Proceed with endotracheal intubation and artificial ventilation at a frequency of 12 times/minute, Vt = 6-8ml/kg, FiO2 50%, I:E = 1:2, PEEP = 5cmH2O, EtCO2 = 35-45mmHg, sevoflurane Install until MAC reaches 0.8-1.
  * Maintain anesthesia with sevofluran, maintain 1 MAC.
  * Using fentanyl during surgery: when ANIm index is less than 50: 50mcg fentanyl bolus, repeat after 5 minutes until ANIm greater than 50. Record the amount of fentanyl used during surgery. Record the ANIm index at the time of the study: when skin incision (T0) and every 10 minutes until the end of surgery.
  * Release of anesthesia: Patients are extubated when they meet the criteria: awake, following orders, breathing rate 12-20 times/minute, SpO2 > 95% with FiO2 ≤ 40%, Vt > 5ml/kg, EtCO2 < 45 mmHg , good cough and swallow reflex and TOF ≥ 90%. After extubation, monitor the patient, record pulse index, blood pressure and VAS score and transfer the patient to the hospital room if it reaches 10/10 points according to Aldrete.
* Pain relief: both groups received paracetamol 1g and ketorolac 30mg at the end of skin closure and every 8 hours thereafter. When the patient has postoperative pain (VAS score ≥ 4), they are titrated with intravenous morphine 1mg/time every 10 minutes until reaching a VAS score < 4. At the same time, an intravenous morphine pain relief machine is installed. Patient controlled analgesia (PCA) with bolus setting 1ml = 1mg, lockout time 10 minutes, maximum dose 20mg/4 hours, no background infusion dose.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I-III.
* Patients had lumbar spinal fusion surgery.

Exclusion Criteria:

* The patient does not agree to participate in the study.
* Patients with severe chronic diseases: liver failure, kidney failure, heart failure, arrhythmia, neuromuscular disease.
* Patients are using drugs that affect the autonomic nervous system such as beta blockers, parasympathomimetic drugs.
* history of mental disorders, difficulty in communication.
* Patients with acute lumbar spine injury or a history of lumbar spine surgery, injections, abscesses, and lumbar infections.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-10-02 (Actual)

PRIMARY OUTCOMES:
The blockade area of TLIP block and ESP block methods | after 20 minutes of block
  Assessing sensory blockade area, according to the pinprick test
The perioperative effectiveness of TLIP block and ESP block methods (aspect 1) | up to the end of surgery
  Evaluating pain relief effectiveness during surgery by total amount of fentanyl used during surgery.
The perioperative effectiveness of TLIP block and ESP block methods (aspect 2) | up to the end of surgery
  Evaluating pain relief effectiveness during surgery by Analgesia Nociception Index (ANIm) scores: ANI is based on electrocardiographic data reflecting parasympathetic activity. ANI creates a value from 0 to 100, where a value greater than 50 indicates adequate analgesia (high parasympathetic tone) and a value less than 50 indicates nociception (a high sympathetic tone) and therefore inadequate analgesia.
The perioperative effectiveness of TLIP block and ESP block methods (aspect 1) | up to 24 hours after extubation
  Evaluating pain relief effectiveness after surgery by total dose of morphine in 12 hours and 24 hours after surgery.
The perioperative effectiveness of TLIP block and ESP block methods (aspect 2) | up to 24 hours after extubation
  Evaluating pain relief effectiveness after surgery by Visual Analogue Scale (VAS) scores at study times within 24 hours after surgery when at rest and on movement (coughing, bending knees). The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').
Side effects | up to 24 hours after extubation
  Rate of vomitting/nausea, itchy, urinary retention, respiratory failure, circulatory failure postoperative of all groups.

CONTACTS AND LOCATIONS:
Overall Officials: Tu Nguyen, Professor, Study Director — Hanoi Medical University
Locations (1):
- Hanoi Medical University, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
The investigators agree that all results and conclusion of this research will be used fully for other researchers
Supporting Information: Study Protocol
Time Frame: from October 2023 to the unidentified time
Access Criteria: anesthesiologists, surgeons all over the world